CLINICAL TRIAL: NCT01767441
Title: Effects of Bariatric Surgeries on Glucose Homeostasis and Its Determinants During a Mixed Meal Tolerance Test
Brief Title: Bariatric Surgeries and Glucose Homeostasis During a Mixed Meal Test
Acronym: BASMEAL
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Sponsor
Other Study IDs: MGZenti MMT
Record Dates: First submitted 2013-01-11; First posted 2013-01-14 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2012-08

CONDITIONS: Obesity
Keywords: bariatric surgery; gastric bypass; gastric banding; sleeve gastrectomy; weight loss; Type 2 Diabetes mellitus; GLP1; obesity; mixed meal test
MeSH Terms: conditions — Obesity; Weight Loss; Diabetes Mellitus, Type 2 | interventions — Gastric Bypass; Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Roux-en-Y-gastric bypass: morbidly obese subjects undergoing gastric bypass surgery
  Interventions: Procedure: Roux-en-Y-gastric bypass
- gastric banding: morbidly obese subjects undergoing laparoscopic adjustable gastric banding
  Interventions: Procedure: laparoscopic adjustable gastric banding
- sleeve gastrectomy: morbidly obese subjects undergoing laparoscopic sleeve gastrectomy
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- control group: morbidly obese subjects not undergoing bariatric surgery, on diet treatment
  Interventions: Other: diet treatment

INTERVENTIONS:
Procedure: Roux-en-Y-gastric bypass — Gastric bypass consisted of creation of a 15-20 ml gastric pouch, a 150 cm Roux limb, and a 50 cm biliopancreatic limb
  Other Names: RYGB
  Groups: Roux-en-Y-gastric bypass
Procedure: laparoscopic adjustable gastric banding — Gastric banding functions by limiting food intake after the placement of an inflatable tube around the stomach just below the gastroesophageal junction, which allows for adjustment of the size of the outlet via the addition or removal of saline through a subcutaneous port.
  Other Names: LAGB
  Groups: gastric banding
Procedure: laparoscopic sleeve gastrectomy — Sleeve gastrectomy involved a gastric reduction of 75 to 80% by resecting the stomach alongside a 30-French endoscope beginning 3 cm from pylorus and ending at the angle of His
  Other Names: SG
  Groups: sleeve gastrectomy
Other: diet treatment — Hypocaloric diet providing a 1000 Kcal/d deficit from total energy expenditure assessed by indirect calorimetry and physical activity determination
  Other Names: diet
  Groups: control group

SUMMARY:
Bariatric surgery can lead to improvement or even resolution of type 2 diabetes Mellitus (T2DM) with the spectrum of responses depending also on operation procedures. However, many mechanisms of metabolic action of different surgical techniques still are unclear.

The aim of this study is to provide a better understanding of the effects of three types of bariatric surgery (lap banding, gastric bypass and sleeve gastrectomy) on beta-cell function and incretin secretion. A mixed meal tolerance (MMT) test will be performed before and 1 and 12 months after surgery to assess beta cell adequacy and glucagon-like-peptide-1 (GLP1)/glucose-dependent insulinotropic polypeptide (GIP) bioavailability.

DETAILED DESCRIPTION:
The effects of different kind of bariatric surgery on glucose homeostasis and its primary determinants (insulin sensitivity and secretion) may differ from one procedure to another. In spite being able to promote improvement/resolution of T2DM, many mechanisms of metabolic action of weight-loss surgery are still unclear. It has been hypothesized that changing the nutrient route through the gut may be a key factor in changing beta cell function and/or insulin sensitivity.

In this study a mixed meal test will be used to assess changes in glucose regulation, beta cell function and incretin bioavailability brought about by different bariatric surgeries in obese patients.

All participants will ingest a standardized mixed meal (163 Kcal; 57% carbohydrate, 33% fat, 22% prot) and will be monitored for 300 minutes thereafter.

Baseline (-20', -10', 0') blood samples will be collected to measure plasma glucose, insulin, C-peptide, incretins and the 13-Carbon-glucose/12-Carbon-glucose (13C-/12C-glucose) ratio (the last one by isotope ratio mass spectrometry).

At time 0', subjects will ingest a standardized mixed meal containing 30 g corn flour and 20 g cheese (parmesan) over 20 minutes. Plasma glucose, insulin, C-peptide, GLP1/GIP and the 13C-/12C-glucose ratio will be assessed at +10', +20', +30', +45', +60', +75', +90', +105', +120', +140', +160', +180', +200', +220', +240', +270', +300'.

Blood samples will be quickly spun at 1500 g at +4°C, plasma/serum will be collected and stored at -80°C.

The 13-Carbon content of maize starch is higher than most of non maize derived sugars. Thus, in individuals on maize and cane sugar free diets, the 13-Carbon/12-Carbon (13C/12C) maize starch ratio is higher (about 10:1000) than the 13C/12C ratio of endogenous glucose derived from glycogenolysis/gluconeogenesis. When these individuals ingest maize starch, the glucose molecules appearing in the systemic circulation which are derived from maize starch will display a 13C-/12C ratio which is identical to maize starch and higher than endogenous glucose. Thus, by measuring the time course of plasma 13C-/12C-glucose ratio, it will be possible to distinguish meal derived glucose from endogenous glucose output (glycogenolysis and gluconeogenesis).

This mixed meal test will be performed before and 1 and 12 months after bariatric surgery. The same tests with the same timing will be performed in a control group of obese patients not undergoing bariatric surgery, being treated with diet only.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 kg/m2.
* BMI ≥ 35 kg/m2 and comorbidities.
* No major organ disease unrelated to excess body weight.
* Mentally able to understand the study and willingness to participate in the study

Exclusion Criteria:

* BMI< 35 kg/m2.
* pregnancy/lactation.
* prior bariatric or gastrointestinal surgery. Malignancies; mental incapacity; unwillingness or language barriers precluding adequate understanding or cooperation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 64 morbidly obese patients will be studied, composed of:
  * 16 subjects scheduled for Roux-en-Y-gastric bypass;
  * 16 subjects scheduled for laparoscopic adjustable gastric banding;
  * 16 subjects scheduled for laparoscopic sleeve gastrectomy;
  * 16 subjects not undergoing bariatric surgery, on diet treatment (control group)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change in glucose response (pAUC) to mixed meal test between baseline and 1 month after undergoing bariatric surgery or being put on low calorie diet | 1 month
  Blood samples will be taken at basal (-20',-10' and 0'), and after the ingestion of a standardized mixed meal (+10', +20', +30',+45', +60', +75', +90', +105', +120', +140', +160', +180', +200', +220', +240', +270', +300').

SECONDARY OUTCOMES:
change in glucose response (pAUC) to mixed meal test between baseline and 12 months after undergoing bariatric surgery or being put on low calorie diet | 12 months
  Blood samples will be taken at basal(-20',-10' and 0'), and after the ingestion of a standardized mixed meal (+10', +20', +30',+45', +60', +75', +90', +105', +120', +140', +160', +180', +200', +220', +240', +270', +300').
changes in β-cell response mixed meal test between baseline and 1 and 12 months after undergoing bariatric surgery or being put on low calorie diet | 1 month and 12 months
  Beta-cell function will be assessed by a state of art mathematical model applied to glucose and C-peptide curves during a standardized mixed meal. Two main metrics of beta cell function will be derived from modeling: 1) derivative or dynamic control of beta cell function, and 2) proportional or static control of beta cell function.
changes in active GLP1 systemic bioavailability during a mixed meal test between baseline and 1 or 12 months after undergoing bariatric surgery or being put on low calorie diet. | 1 month and 12 months
  Blood samples will be taken at basal(-20',-10' and 0'), and after the ingestion of a standardized mixed meal (+10', +20', +30',+45', +60', +75', +90', +105', +120', +140', +160', +180', +200', +220', +240', +270', +300').

OTHER OUTCOMES:
change in HbA1c between baseline and 1 or 12 months after undergoing bariatric surgery or being put on low calorie diet. | 1 month and 12 months
  high pressure liquid chromatography (HPLC) method

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Zenti, MD, Principal Investigator — Division of Endocrinology and Metabolic Diseases, AOUI Verona, Italy; Enzo Bonora, Professor, Study Director — Division of Endocrinology and Metabolic Diseases, University Hospital of Verona
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No